CLINICAL TRIAL: NCT04047420
Title: A Phase 1 Open Label Safety and Pharmacokinetic Study of Rectal Administration of a Tenofovir Alafenamide/Elvitegravir Insert at Two Dose Levels
Brief Title: Safety and Pharmacokinetic Study of Tenofovir Alafenamide (TAF)/Elvitegravir (EVG) Administered Rectally
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MTN-039; 38470 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tenofovir Alafenamide (TAF)/Elvitegravir (EVG) Insert (Experimental): On the first dosing visit (Visit 3), participants will receive a single TAF/EVG Insert for rectal administration. On the second dosing visit (Visit 7), after a washout period of at least 7 days, participants will receive two TAF/EVG Inserts for rectal administration. Each participant will be on study for approximately 6-13 weeks.
  Interventions: Drug: TAF/EVG Insert

INTERVENTIONS:
Drug: TAF/EVG Insert — TAF/EVG Insert (20/16 mg) administered rectally by study staff

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of rectal administration of a tenofovir alafenamide (TAF)/elvitegravir (EVG) insert at two dose levels in HIV-uninfected individuals.

DETAILED DESCRIPTION:
This study will evaluate the safety and pharmacokinetics of rectal administration of a tenofovir alafenamide (TAF)/elvitegravir (EVG) insert at two dose levels in HIV-uninfected individuals.

All participants will receive a single TAF/EVG Insert at Study Visit 3. After a washout period of at least 7 days, participants will receive two TAF/EVG Inserts at Study Visit 7. The inserts will be administered rectally by study staff. After each dosing visit, samples will be collected over a 3-day period.

Participants will attend 10 study visits and will be followed for approximately 6 to 13 weeks. Study visits may include physical and rectal examinations; collection of blood, urine, rectal and vaginal fluid; and interviews. The total duration of the study will be approximately 11 months.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are 18 years of age or older at Screening, verified per site standard operating procedure (SOP)
* Able and willing to provide written informed consent to be screened for and enrolled in MTN-039
* HIV-1/2 uninfected at Screening and Enrollment, per applicable algorithm in the study protocol and willing to receive HIV test results
* Able and willing to provide adequate locator information, as defined in site SOP
* Able to communicate in spoken and written English
* Available for all visits and able and willing to comply with all study procedural requirements
* In general good health at Screening and Enrollment, as determined by the site Investigator of Record (IoR) or designee
* At Screening, history of consensual receptive anal intercourse (RAI) at least once in lifetime per participant report
* Willing not to take part in other research studies involving drugs, medical devices, genital or rectal products, or vaccines for the duration of study participation (including the time between Screening and Enrollment)
* Willing to comply with abstinence and other protocol requirements as outlined in the study protocol
* For participants of childbearing potential: a negative pregnancy test at Screening and Enrollment
* For participants of childbearing potential: Per participant report at Enrollment, using an effective method of contraception for at least 30 days (inclusive) prior to Enrollment and intending to use an effective method for the duration of study participation. Effective methods include:

  * Hormonal methods
  * Intrauterine device (IUD) inserted at least 30 days prior to Enrollment (but not past the maximum length of recommended usage according to package instructions)
  * Sterilization (of participant or partner, as defined in site SOPs)
  * Sexually abstinent as defined by abstaining from penile-vaginal intercourse for 90 days prior to Enrollment and intending to remain abstinent for the duration of study participation; this includes having sex exclusively with individuals assigned female sex at birth

Exclusion Criteria:

* At Screening:

  * Hemoglobin Grade 1 or higher*
  * Platelet count Grade 1 or higher*
  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) Grade 1 or higher*
  * Serum creatinine greater than 1.3 times the site laboratory upper limit of normal (ULN)
  * International normalized ratio (INR) greater than 1.5 times the site laboratory ULN
  * History of inflammatory bowel disease by participant report
  * Positive hepatitis B surface antigen (HBsAg) test result
  * *As per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1, July 2017.
  * Note: Otherwise eligible participants with an exclusionary test result (other than HIV) can be re-tested during the screening process. If a participant is re-tested and a non-exclusionary result is documented within 45 days of providing informed consent for screening, the participant may be enrolled.
* Anticipated use of and/or unwillingness to abstain from the following medications during study participation:

  * Anticoagulant medications
  * Non-study rectally-administered medications and any products containing nonoxynol-9 (N-9)
* Known adverse reaction to any of the components of the study product
* Use of approved or other investigational pre-exposure prophylaxis (PrEP) for HIV prevention within 3 months prior to Enrollment, and/or anticipated use and/or unwillingness to abstain from PrEP during trial participation
* Use of post-exposure prophylaxis (PEP) for potential HIV exposure within 6 months prior to Enrollment
* Condomless RAI and/or penile-vaginal intercourse with a partner who is known to be HIV-positive or whose status is unknown in the 6 months prior to Enrollment
* History of transactional sex in the 12 months prior to Enrollment
* Non-therapeutic injection drug use or use of non-therapeutic, non-injection stimulant drugs in the 12 months prior to Enrollment
* Participation in research studies involving drugs, medical devices, genital or rectal products, or vaccines within 30 days of the Enrollment Visit
* Per participant report, medical records, clinical diagnosis and/or diagnostic testing at either Screening or Enrollment:

  * Diagnosis or treatment of an anogenital sexually transmitted infection (STI) in the 3 months prior to enrollment (including window between Screening and Enrollment).
  * Symptoms, clinical or laboratory diagnosis of active pharyngeal, anorectal, or reproductive tract infection (RTI) requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines (http://www.cdc.gov/std/treatment).
  * Current symptomatic urinary tract infection (UTI).

    * Infections requiring treatment include Neisseria gonorrhea (GC), Chlamydia trachomatis (CT) infection, syphilis, active herpes simplex virus (HSV) lesions, or symptomatic genital warts, chancroid, pelvic inflammatory disease (PID), bacterial vaginosis (BV), symptomatic vaginal candidiasis, and trichomoniasis.
    * Note: Otherwise eligible participants with an exclusionary UTI, BV and/or candida finding may be re-tested during the screening process.
* For participants of childbearing potential: Pregnant or breastfeeding at either Screening or Enrollment or planning to become pregnant during study participation

  * Note: A documented negative pregnancy test performed by study staff is required for inclusion; however, a self-reported pregnancy is adequate for exclusion from screening/enrollment into the study.
* For participants of childbearing potential: Last pregnancy outcome 90 days or less prior to Screening
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate the interpretation of study outcome data, or otherwise interfere with achieving the study objectives including any significant uncontrolled active or chronic medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A. Riddler, MD, MPH, Study Chair — University of Pittsburgh
Locations (2):
- United States (2):
  - Alabama CRS, Birmingham, Alabama
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Riddler SA, Kelly CW, Hoesley CJ, Ho KS, Piper JM, Edick S, Heard F, Doncel GF, Johnson S, Anderson PL, Brand RM, Kunjara Na Ayudhya RP, Bauermeister JA, Hillier SL, Hendrix CW. A Phase 1 Clinical Trial to Assess the Safety and Pharmacokinetics of a Tenofovir Alafenamide/Elvitegravir Insert Administered Rectally for HIV Prevention. J Infect Dis. 2024 Sep 23;230(3):696-705. doi: 10.1093/infdis/jiae211. PMID 38655842

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 23 participants were eligible and enrolled. Two participants terminated early due to "Refused participation", so 21 participants received the one insert dose. After the one insert dose, two additional participants terminated early due to "Refused participation", so 19 participants received the two insert dose.
Period: Enrollment (Pre-dose) Period
Arm/Group | Tenofovir Alafenamide (TAF)/Elvitegravir (EVG) Insert
Started | 23
Completed | 21
Not Completed | 2
Not completed — Refused Participation | 2
Period: One TAF/EVG Insert Dose
Arm/Group | Tenofovir Alafenamide (TAF)/Elvitegravir (EVG) Insert
Started | 21
Completed | 21
Not Completed | 0
Period: Washout Period
Arm/Group | Tenofovir Alafenamide (TAF)/Elvitegravir (EVG) Insert
Started | 21
Completed | 19
Not Completed | 2
Not completed — Refused Participation | 2
Period: Two TAF/EVG Inserts Dose
Arm/Group | Tenofovir Alafenamide (TAF)/Elvitegravir (EVG) Insert
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tenofovir Alafenamide (TAF)/Elvitegravir (EVG) Insert
Number analyzed (Participants) | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.0 [24 to 43]
Age, Customized [Count of Participants; unit: Participants]
  24 years or Under | 6
  25-29 years | 2
  30-34 years | 4
  35-39 years | 3
  40-44 years | 4
  45-49 years | 1
  50+ years | 3
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 15
  Gender: Female | 6
  Gender: Transgender Male | 0
  Gender: Transgender Female | 1
  Gender: Gender Nonconforming/Gender Variant | 0
  Gender: Self-identify | 0
  Gender: Prefer Not to Answer | 0
  Gender: Multiple Genders | 1
Sex: Female, Male [Count of Participants; unit: Participants] — at birth
  Participants
    Female | 17
    Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 0
  Race: Black or African American | 8
  Race: Native Hawaiian or other Pacific Islander | 0
  Race: White | 13
  Race: Other | 1
  Race: Mixed | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Pittsburgh | 11
  United States: Birmingham | 12
Sexual Orientation [Count of Participants; unit: Participants]
  Gay/Lesbian/Homosexual | 11
  Bisexual | 6
  Queer | 0
  Two Spirit | 0
  Straight/Heterosexual | 5
  Additional Category | 1
  Not sure | 0
  Prefer not to Answer | 0
Participant Height (cm) [Median (Inter-Quartile Range); unit: cm] | 175.0 [166 to 182]
Participant Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 93.0 [75 to 116]
Participant BMI (kg/m^2) [Median (Inter-Quartile Range); unit: kg/m^2] | 30.8 [26 to 37]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 2 and Higher Adverse Events (AEs)
Description: Graded per the Division of AIDS (DAIDS) Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 and/or Addenda 1, 2 and 3 (Female Genital [Dated November 2007], Male Genital [Dated November 2007] and Rectal [Clarification Dated May 2012] Grading Tables for Use in Microbicide Studies).
Time Frame: Measured from Enrollment through Final Contact at Visit 11 with a median (IQR) of 76 (47, 292) days. COVID restrictions delayed first dosing 9-10 months in 5 participants. Follow-up time from first dosing was a median (IQR) of 34 (22, 39) days.
Population: All participants with dosing of one insert or two inserts.
Measure: Count of Participants; unit: Participants
Groups:
- One Insert: All participants who received a single TAF/EVG rectal insert
- Two Inserts: All participants who received two TAF/EVG rectal inserts
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
Participants
  Participants experiencing grade 2+ AE: Yes | 1 | 1
  Participants experiencing grade 2+ AE: No | 20 | 18
  Gastritis: Yes | 0 | 1
  Gastritis: No | 21 | 18
  Reactogenicity event: Yes | 1 | 0
  Reactogenicity event: No | 20 | 19

2. Primary Outcome: Elvitegravir (EVG) Concentration in Blood
Description: Based on laboratory evaluations on samples collected at baseline (pre dose), 1, 2, 4, 6, 24, 48, and 72 hours post dose
Time Frame: Samples collected at baseline (pre dose), 1, 2, 4, 6, 24, 48, and 72 hours after each dose (up to 9 weeks after first dose)
Population: Baseline data were collected once at the enrollment visit prior to receiving both one insert and two inserts.
  Participants had post dose blood samples collected at 1, 2, 4, 6, 24, 48, and 72 hours (One insert (n=21); Two inserts (n=19))).
  Missed sample collection (One insert (24-hour missed (n=1)); Two inserts (48-hour missed (n=1) and 72-hour missed (n=1))).
  Unable to draw sample (One insert (72-hours (n=1))).
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
pg/mL
  Baseline (Enrollment Visit): number analyzed (Participants) | 21 | 0
  Baseline (Enrollment Visit) | NA [NA to NA] — Below the Limit of Quantification |
  1 hour postdosing | 1010.0 [564.0 to 2050.0] | 1510.0 [812.0 to 1890.0]
  2 hours postdosing | 1230 [605.0 to 3090.0] | 2140.0 [1240.0 to 3420.0]
  4 hours postdosing | 1080.0 [450.0 to 1960.0] | 1740.0 [933.0 to 3560.0]
  6 hours postdosing | 713.0 [441.0 to 1730.0] | 1290.0 [825.0 to 2230.0]
  24 hours postdosing: number analyzed (Participants) | 20 | 19
  24 hours postdosing | 39.0 [NA to 201.5] — Below the Limit of Quantification | 76.0 [35.0 to 471.0]
  48 hours postdosing: number analyzed (Participants) | 21 | 18
  48 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification
  72 hours postdosing: number analyzed (Participants) | 20 | 18
  72 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification

3. Primary Outcome: Elvitegravir (EVG) Concentration in Rectal Fluid
Description: Based on laboratory evaluations on samples collected at 2, 4, 6, 24, 48, and 72 hours post dose
Time Frame: Samples collected at 2, 4, 6, 24, 48, and 72 hours after each dose (up to 9 weeks after first dose)
Population: Participants are randomly assigned 1:1 to post dose rectal fluid sampling at either 2, 6, and 48 hours (One insert (n=10); Two inserts (n=9)) or 4, 24, and 72 hours (One insert (n=11); Two inserts (n=10)).
  Missed sample collection (One insert (24-hour missed (n=1) but replaced by 48-hour sample); Two inserts (48-hour missed (n=1))).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
ng/mL
  2 hours postdosing: number analyzed (Participants) | 10 | 9
  2 hours postdosing | 67542.0 [31652.0 to 338721.0] | 176672.0 [50962.0 to 731606.0]
  4 hours postdosing: number analyzed (Participants) | 11 | 10
  4 hours postdosing | 125676.0 [72779.0 to 319693.0] | 93888.5 [49922.0 to 236267.0]
  6 hours postdosing: number analyzed (Participants) | 10 | 9
  6 hours postdosing | 4095.5 [338.0 to 8708.0] | 7791.0 [619.0 to 13131.0]
  24 hours postdosing: number analyzed (Participants) | 10 | 10
  24 hours postdosing | 2233.5 [574.0 to 3517.0] | 2596.5 [89.1 to 18664.0]
  48 hours postdosing: number analyzed (Participants) | 11 | 8
  48 hours postdosing | 16.9 [2.1 to 278.0] | 36.4 [1.0 to 807.5]
  72 hours postdosing: number analyzed (Participants) | 11 | 10
  72 hours postdosing | 5.9 [NA to 16.5] — Below the Limit of Quantification | 29.1 [2.3 to 58.1]

4. Primary Outcome: Elvitegravir (EVG) Concentration in Rectal Mucosal Tissue Homogenates
Description: Based on laboratory evaluations on samples collected at 2, 24, 48, and 72 hours post dose
Time Frame: Samples collected at 2, 24, 48, and 72 hours after each dose (up to 9 weeks after first dose)
Population: Participants are randomly assigned 1:1 to post dose rectal tissue sampling at either 2 and 48 hours (One insert (n=10)); Two inserts (n=9)) or 24 and 72 hours (One insert (n=11); Two inserts (n=10)).
  Missed sample collection (One insert (24-hour missed (n=1)); Two inserts (48-hour missed (n=1) and 72-hour missed (n=1))).
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
ng/mg
  2 hours postdosing: number analyzed (Participants) | 10 | 9
  2 hours postdosing | 5.4 [0.6 to 10.2] | 9.0 [5.3 to 35.3]
  24 hours postdosing: number analyzed (Participants) | 10 | 10
  24 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | 0.1 [NA to 0.7] — Below the Limit of Quantification
  48 hours postdosing: number analyzed (Participants) | 10 | 8
  48 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification
  72 hours postdosing: number analyzed (Participants) | 11 | 9
  72 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification

5. Primary Outcome: Tenofovir Alafenamide (TAF) Concentration in Blood
Description: Based on laboratory evaluations on samples collected at baseline (pre dose), 1, 2, 4, 6, 24, 48, and 72 hours post dose
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
pg/mL
  Baseline (Enrollment visit): number analyzed (Participants) | 21 | 0
  Baseline (Enrollment visit) | NA [NA to NA] — Below the Limit of Quantification |
  1 hour postdosing | 29500.0 [16700.0 to 37900.0] | 40400.0 [22600.0 to 65900.0]
  2 hours postdosing | 14000.0 [5850.0 to 32100.0] | 26200.0 [8970.0 to 54300.0]
  4 hours postdosing | 747.0 [169.0 to 1660.0] | 1350.0 [525.0 to 6650.0]
  6 hours postdosing | 56.0 [NA to 222.0] — Below the Limit of Quantification | 95.0 [27.0 to 427.0]
  24 hours postdosing: number analyzed (Participants) | 20 | 19
  24 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification
  48 hours postdosing: number analyzed (Participants) | 21 | 18
  48 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification
  72 hours postdosing: number analyzed (Participants) | 20 | 18
  72 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification

6. Primary Outcome: Tenofovir Alafenamide (TAF) Concentration in Rectal Fluid
Description: Based on laboratory evaluations on samples collected at 2, 4, 6, 24, 48, and 72 hours post dose
Time Frame: Samples collected at 2, 4, 6, 24, 48, and 72 hours after each dose (up to 9 weeks after first dose)
Population: Participants are randomly assigned 1:1 to post dose rectal fluid sampling at either 2, 6, and 48 hours (One insert (n=10); Two inserts (n=9)) or 4, 24, and 72 hours (One insert (n=11); Two inserts (n=10)).
  Missed sample collection (One insert (24-hour missed (n=1) but replaced by 48-hour sample); Two inserts (48-hour missed (n=1))).
  Rejected samples, no results (One insert (2-hours (n=1), 4-hours (n=2), and 6-hours (n=2)); Two inserts (6-hours (n=1) and 48-hours (n=1))).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
ng/mL
  2 hours postdosing: number analyzed (Participants) | 9 | 9
  2 hours postdosing | 1394.0 [358.0 to 6085.0] | 531.0 [196.0 to 16080.0]
  4 hours postdosing: number analyzed (Participants) | 9 | 10
  4 hours postdosing | 1279.0 [53.7 to 6056.0] | 954.0 [308.0 to 6008.0]
  6 hours postdosing: number analyzed (Participants) | 8 | 8
  6 hours postdosing | 10.8 [1.2 to 30.1] | 12.4 [1.3 to 58.4]
  24 hours postdosing: number analyzed (Participants) | 10 | 10
  24 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | 0.6 [NA to 3.9] — Below the Limit of Quantification
  48 hours postdosing: number analyzed (Participants) | 11 | 7
  48 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification
  72 hours postdosing: number analyzed (Participants) | 11 | 10
  72 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification

7. Primary Outcome: Tenofovir Alafenamide (TAF) Concentration in Rectal Mucosal Tissue Homogenates
Description: Based on laboratory evaluations on samples collected at 2, 24, 48, and 72 hours post dose
Time Frame: Samples collected at 2, 24, 48, and 72 hours after each dose (up to 9 weeks after first dose)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
ng/mg
  2 hours postdosing: number analyzed (Participants) | 10 | 9
  2 hours postdosing | NA [NA to 0.1] — Below the Limit of Quantification | NA [NA to 0.1] — Below the Limit of Quantification
  24 hours postdosing: number analyzed (Participants) | 10 | 10
  24 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification
  48 hours postdosing: number analyzed (Participants) | 10 | 8
  48 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification
  72 hours postdosing: number analyzed (Participants) | 11 | 9
  72 hours postdosing | NA [NA to NA] — Below the Limit of Quantification | NA [NA to NA] — Below the Limit of Quantification

8. Primary Outcome: Tenofovir (TFV) Concentration in Blood
Description: Based on laboratory evaluations on samples collected at baseline (pre dose), 1, 2, 4, 6, 24, 48, and 72 hours post dose
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
pg/mL
  Baseline (Enrollment visit): number analyzed (Participants) | 21 | 0
  Baseline (Enrollment visit) | NA [NA to NA] — Below the Limit of Quantification |
  1 hour postdosing | 1290.0 [796.0 to 1880.0] | 2140.0 [1520.0 to 3070.0]
  2 hours postdosing | 2080.0 [1690.0 to 3430.0] | 3700.0 [2490.0 to 5170.0]
  4 hours postdosing | 2380.0 [1510.0 to 3580.0] | 4080.0 [2360.0 to 5520.0]
  6 hours postdosing | 1780.0 [1050.0 to 3010.0] | 3420.0 [1910.0 to 4640.0]
  24 hours postdosing: number analyzed (Participants) | 20 | 19
  24 hours postdosing | 1105.0 [558.5 to 1995.0] | 1910.0 [1100.0 to 3210.0]
  48 hours postdosing: number analyzed (Participants) | 21 | 18
  48 hours postdosing | 570.0 [311.0 to 1020.0] | 1085.0 [852.0 to 1480.0]
  72 hours postdosing: number analyzed (Participants) | 20 | 18
  72 hours postdosing | 340.5 [133.0 to 696.0] | 687.0 [438.0 to 841.0]

9. Primary Outcome: Tenofovir (TFV) Concentration in Rectal Fluid
Description: Based on laboratory evaluations on samples collected at 2, 4, 6, 24, 48, and 72 hours post dose
Time Frame: Samples collected at 2, 4, 6, 24, 48, and 72 hours after each dose (up to 9 weeks after first dose)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
ng/mL
  2 hours postdosing: number analyzed (Participants) | 9 | 9
  2 hours postdosing | 18086.0 [15509.0 to 34292.0] | 43188.0 [26667.0 to 78240.0]
  4 hours post dosing: number analyzed (Participants) | 9 | 10
  4 hours post dosing | 85434.0 [37836.0 to 126430.0] | 100834.5 [58003.0 to 141675.0]
  6 hours postdosing: number analyzed (Participants) | 8 | 8
  6 hours postdosing | 9794.0 [2076.5 to 18268.0] | 10214.5 [5255.0 to 26800.5]
  24 hours postdosing: number analyzed (Participants) | 10 | 10
  24 hours postdosing | 2909.0 [1744.0 to 8465.0] | 8276.5 [5261.0 to 23540.0]
  48 hours postdosing: number analyzed (Participants) | 11 | 7
  48 hours postdosing | 924.0 [337.0 to 2010.0] | 1057.0 [687.0 to 2289.0]
  72 hours postdosing: number analyzed (Participants) | 11 | 10
  72 hours postdosing | 380.0 [41.8 to 881.0] | 545.5 [78.2 to 1011.0]

10. Primary Outcome: Tenofovir (TFV) Concentration in Rectal Mucosal Tissue Homogenates
Description: Based on laboratory evaluations on samples collected at 2, 24, 48, and 72 hours post dose
Time Frame: Samples collected at 2, 24, 48, and 72 hours after each dose (up to 9 weeks after first dose)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
ng/mg
  2 hours postdosing: number analyzed (Participants) | 10 | 9
  2 hours postdosing | 15.4 [3.2 to 35.6] | 28.4 [16.7 to 40.6]
  24 hours postdosing: number analyzed (Participants) | 10 | 10
  24 hours postdosing | 1.5 [0.2 to 9.8] | 10.2 [2.5 to 21.9]
  48 hours postdosing: number analyzed (Participants) | 10 | 8
  48 hours postdosing | 2.3 [NA to 5.1] — Below the Limit of Quantification | 3.3 [2.3 to 5.5]
  72 hours postdosing: number analyzed (Participants) | 11 | 9
  72 hours postdosing | NA [NA to 2.1] — Below the Limit of Quantification | 1.0 [0.4 to 5.2]

11. Primary Outcome: Tenofovir Diphosphate (TFV-DP) Concentration in Rectal Mucosal Tissue Cell Isolates
Description: Based on laboratory evaluations on samples collected at 2, 24, 48, and 72 hours post dose
Time Frame: Samples collected at 2, 24, 48, and 72 hours after each dose (up to 9 weeks after first dose)
Population: Participants are randomly assigned 1:1 to post dose rectal tissue sampling at either 2 and 48 hours (One insert (n=10)); Two inserts (n=9)) or 24 and 72 hours (One insert (n=11); Two inserts (n=10)).
  Missed sample collection (One insert (24-hour missed (n=1)); Two inserts (48-hour missed (n=1) and 72-hour missed (n=1))).
  Rejected samples, no results (One insert (2-hours (n=2) and 48-hours (n=2)); Two inserts (48-hours (n=1) and 72-hours (n=1))).
Measure: Median (Inter-Quartile Range); unit: fmol/10^6 Cells
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
fmol/10^6 Cells
  2 hours postdosing: number analyzed (Participants) | 8 | 9
  2 hours postdosing | 8219.0 [3443.0 to 12723.0] | 6230.0 [5704.0 to 12783.0]
  24 hours postdosing: number analyzed (Participants) | 10 | 10
  24 hours postdosing | 2315.5 [335.0 to 8055.0] | 6727.0 [2189.0 to 12295.0]
  48 hours postdosing: number analyzed (Participants) | 8 | 7
  48 hours postdosing | 2459.0 [89.0 to 4559.0] | 2822.0 [815.0 to 3599.0]
  72 hours postdosing: number analyzed (Participants) | 11 | 8
  72 hours postdosing | 149.0 [43.6 to 1075.0] | 2022.0 [347.0 to 3122.0]

12. Secondary Outcome: Participant Self-report Rectal Insert Acceptability - Ease of Use
Description: Response for "Overall, how easy or difficult was it to use the study product when inserted by clinic staff?
Time Frame: 24 hours after each dose (Visits 4 and 8) (up to 9 weeks after first dose)
Population: All participants who completed the follow-up computer-administered self-interview (CASI) questionnaire at 24 hours post-dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
Participants
  Very difficult | 0 | 0
  Difficult | 0 | 0
  Easy | 7 | 8
  Very easy | 14 | 11
  Decline to answer | 0 | 0

13. Secondary Outcome: Participant Self-report Rectal Insert Acceptability - Feeling When Inserted
Description: Response for "How did it feel to have the insert inside you?"
Time Frame: 24 hours after each dose (Visits 4 and 8) (up to 9 weeks after first dose)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
Participants
  Very comfortable | 8 | 8
  Comfortable | 10 | 10
  Uncomfortable | 2 | 1
  Very uncomfortable | 0 | 0
  Decline to answer | 1 | 0

14. Secondary Outcome: Participant Self-report Rectal Insert Acceptability - Problems With Rectal Insert
Description: Responses for questions related to problems with Rectal Insert
Time Frame: 24 hours after each dose (Visits 4 and 8) (up to 9 weeks after first dose)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | One Insert | Two Inserts
Number analyzed (Participants) | 21 | 19
Participants
  Did you have any problems using the study insert after it was inserted?: No | 20 | 19
  Did you have any problems using the study insert after it was inserted?: Yes | 1 | 0
  Did you have any problems using the study insert after it was inserted?: Decline to answer | 0 | 0
  Did you experience any leakage after you used the insert?: No | 20 | 18
  Did you experience any leakage after you used the insert?: Yes | 1 | 1
  Did you experience any leakage after you used the insert?: Decline to answer | 0 | 0
  Since your last study visit, have you experienced any soiling of your underwear or linens?: No | 20 | 18
  Since your last study visit, have you experienced any soiling of your underwear or linens?: Yes | 1 | 1
  Since your last study visit, have you experienced any soiling of your underwear or linens?: Decline to answer | 0 | 0
  Since your last study visit, have you experienced any diarrhea?: No | 20 | 18
  Since your last study visit, have you experienced any diarrhea?: Yes | 1 | 1
  Since your last study visit, have you experienced any diarrhea?: Decline to answer | 0 | 0
  Since your last visit, have you experienced any other stomach or abdominal problems?: No | 12 | 9
  Since your last visit, have you experienced any other stomach or abdominal problems?: Yes | 9 | 10
  Since your last visit, have you experienced any other stomach or abdominal problems?: Decline to answer | 0 | 0

ADVERSE EVENTS:
Time Frame: Measured from Enrollment through Final Contact at Visit 11 with a median (IQR) of 76 (47, 292) days. COVID restrictions delayed first dosing 9-10 months in 5 participants. Follow-up time from first dosing was a median (IQR) of 34 (22, 39) days.
Description: COVID-19 pandemic related scheduling delays occurred for seven participants resulting in collection of pre-dose adverse events over a 9-10 month period prior to first dosing. Of the 23 participants enrolled, two of these seven participants did not return for first dosing, thus 21 participants received the one insert dose.
Groups:
- Baseline (Pre-dosing): All participants who were enrolled in the study, prior to any inserts.
Arm/Group | Baseline (Pre-dosing) | One Insert | Two Inserts
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 3/23 | 4/21 | 4/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline (Pre-dosing) (N=23) | One Insert (N=21) | Two Inserts (N=19)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Reactogenicity event (General disorders) | 1 (1) | 2 (2) | 1 (1) — reactogenicity symptoms
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — right shoulder pain
Urinary tract infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — extrapyramidal symptoms
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — rectal erythema
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Perianal tear
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — Minor vaginal discomfort
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Diarrhea
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT04047420/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT04047420/SAP_001.pdf